CLINICAL TRIAL: NCT04795635
Title: A Prospective, Randomized, Clinical Trial Comparing the Safety and Effectiveness of Axon Therapy for Post-Traumatic Peripheral Neuropathic Pain (PTPNP) to Conventional Medical Management (CMM)
Brief Title: Axon Therapy for Post-Traumatic Peripheral Neuropathic Pain Compared to Conventional Medical Management
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NeuraLace Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NLM-001
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Neuropathic Pain; Peripheral Neuropathy
Keywords: transcutaneous magnetic stimulation; axon therapy; post-traumatic peripheral neuropathic pain
MeSH Terms: conditions — Neuralgia; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled, multi-center, clinical trial in which 80 participants diagnosed with PTPNP will be randomized 1:1 into one of two treatment groups:
  1. CMM plus Axon Therapy (n=64)
  2. CMM alone (n=64)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CMM + Axon Therapy (Experimental): Participants will return to the clinic for assessment at Day 30 (± 14 days), Day 90 (± 14 days), Day 180 (± 30 days) and Day 365 (± 30 days). Participants randomized to the CMM plus Axon Therapy group will return to the clinic for Axon Therapy treatments as follows:
  * Month 1: 6 treatments
    * WEEK 1: 3 treatments (consecutive treatments are best)
    * WEEK 2-4: Weekly treatments
  * Month 2: Bi-monthly treatment
  * Months 3-12: Treatments every 2-4 weeks
  In addition to in-clinic assessments and treatments, all participants will a receive weekly phone follow-up to assess pain intensity and occurrence of adverse events after treatment starts. Weekly phone follow-ups will only occur during weeks when the participant is not in clinic for treatment.
  Interventions: Device: CMM + Axon Therapy
- CMM Only (No Intervention): Participants will return to the clinic for assessment at Day 30 (± 14 days), Day 90 (± 14 days), Day 180 (± 30 days) and Day 365 (± 30 days)

INTERVENTIONS:
Device: CMM + Axon Therapy — transcutaneous magnetic stimulation (tMS)
  Arms: CMM + Axon Therapy

SUMMARY:
Compare Axon Therapy using transcutaneous magnetic stimulation (tMS) against conventional medical management in treating post-traumatic peripheral neuropathic pain (PTPNP).

DETAILED DESCRIPTION:
Subjects will be consented, screened, and undergo a 7-day baseline assessment to measure pain scores and assess diary compliance. Subjects who meet inclusion criteria will undergo an in-clinic baseline evaluation, receive randomization assignment, and start their respective treatments.

Those randomized to the CMM plus Axon Therapy group will receive their first Axon Therapy treatment and then have a follow-up phone call after 24 hours to assess if the patient is a candidate for Axon Therapy, that is if the subject is neuropathic or nociceptive. Those that are not candidates for Axon Therapy will be monitored for 30 days for AEs and then they will exit the study as screen failures. Screen failures will not count against enrollment numbers.

All subjects will return to the clinic for follow-up assessment at Day 30 (± 14 days), Day 90 (± 14 days), Day 180 (± 14 days) and Day 365 (± 30 days) and if in the CMM plus Axon Therapy group will return to the clinic for Axon Therapy treatments as follows:

* Month 1: 6 treatments

  * WEEK 1: 3 treatments (consecutive treatments are best)
  * WEEK 2-4: Weekly treatments
* Month 2: Bi-Weekly treatment
* Months 3-12: Treatments every 2-4 weeks
* Additional treatments to treat flare ups; defined as an episode of pain with a VAS >greater or equal to 6 following an increase in daily activities.

At day 90 (± 15 days), subjects will be allowed to crossover to the alternative treatment group. Subjects who crossover from CMM to CMM plus Axon Therapy will follow the CMM plus Axon Therapy regimen, remaining in the study for 15 months. These subjects will have follow-up visits at Day 120 (± 14 days), Day 180 (± 14 days) ,Day 270 (± 14 days), and Day 450 (± 30 days).

Subjects who crossover from CMM plus Axon Therapy to CMM will be monitored for 30 days for AEs and then they will exit the study. The reason for ending therapy will be recorded.

In addition to in-clinic assessments and treatments, all subjects will complete an electronic daily diary up to twice daily throughout the first 90 days and for crossover subjects they will complete 90 days of Axon treatment therapy and up to Day 180. They will receive weekly phone follow-up to assess pain intensity and occurrence of adverse events after treatment starts. Weekly phone follow-ups will only occur during weeks when the subject is not seen in the clinic.

ELIGIBILITY:
Inclusion Criteria

1. Evidence of a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the study.
2. Subject is willing and able to comply with scheduled visits, treatment plan, daily pain, and other study procedures subject is able and willing to complete twice daily diary.
3. Subject must be literate in English to fill out the study questionnaires.
4. Men or women of any race or ethnicity who are 18-75 years of age.
5. Subject must have chronic peripheral neuropathic pain present for more than three months after a traumatic or surgical event per medical history (this may include, for example, motor vehicle accident, fall, sports injury, knee or hip replacement, hernia repair, thoracotomy, mastectomy, focal/localized burns, or crush injury).
6. Subject has a score ≥6 on VAS at Enrollment/Screening Visit.
7. Subject has completed at least one of the two daily pain diary entries on at least three days between the Enrollment/Screening Visit and Randomization Visit (Visit 1) with a mean pain score of ≥4 and ≤10 based on Daily VAS to be eligible for randomization.
8. Subject has been on a stable pain medication regimen for at least 28 days or is not taking pain medications, as determined by the investigator, at the baseline assessment in this study.
9. Subject must have their implicated peripheral nerve(s) identified and documented in their medical record.

Exclusion Criteria

1. Subjects with neuropathic pain due to post-herpetic neuropathy, HIV, trigeminal neuralgia, or carpal tunnel syndrome; subjects whose post- traumatic neuropathic pain is categorized as central (e.g., spinal cord injury) rather than peripheral.
2. Subject has a currently diagnosed progressive neurological disease such as multiple sclerosis, chronic inflammatory demyelinating polyneuropathy, rapidly progressive arachnoiditis, brain or spinal cord tumor, or severe/critical spinal stenosis (stenosis).
3. Subjects with skin conditions in the affected dermatome that in the judgment of the investigator could interfere with evaluation of the neuropathic pain condition.
4. Subjects with other pain that may confound assessment or self-evaluation of the peripheral neuropathic pain; subjects with significant somatic pain at the site of their trauma that may confound assessment or self-evaluation of their neuropathic pain.
5. Participation in any other clinical trial within the 30 days prior to screening and/or during participation in this study.
6. Any subject considered at risk of suicide or self-harm based on investigator judgment and/or the details of a risk assessment.
7. Other severe acute or chronic medical or psychiatric conditions, or laboratory abnormality, or other factors that may increase the risk associated with study participation or investigational product administration or may interfere with compliance or the interpretation of study results and, in the judgment of the investigator would make the subject inappropriate to participate in the study.
8. Subjects with pending Worker's Compensation, Worker's Compensation, civil litigation, or disability claims pertinent to the subject based upon trauma; current involvement in out-of-court settlements for claims pertinent to subject's trauma; Subjects with fully resolved litigation and compensation claims can participate.
9. Subjects who have had a diagnosis of malignancy other than basal cell carcinoma, or carcinoma in situ of the cervix within the past five years, to include life expectancy less than 1 year due to advanced malignancy.
10. Subjects with implantable "electrical" medical devices such as a cardiac pacemaker, defibrillator, or insulin pump within four (4) inches or less of the site of pain to be treated by Axon Therapy. (Subject with an implantable device greater than four (4) inches from the site of pain to be treated should NOT be excluded).
11. Phantom limb pain or pain that feels like it is coming from a body part that is no longer there.
12. Subjects who have failed other neuromodulation implantable device for the same indication
13. Subjects with shrapnel or ferromagnetic objects
14. Subject is currently taking a morphine equivalent daily dose > 120 mg/day.
15. Subject is a woman of childbearing potential, not using adequate contraception as per investigator judgment or not willing to comply with contraception for the duration of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-08-22 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Proportion of Responders | 90 days
  The primary effectiveness endpoint is a between groups comparison of the proportion of responders, defined as a subject who experiences 50% or greater reduction from baseline in neuropathic pain intensity as measured by in-clinic visual analog score (VAS) for primary area of pain at Day 90 with no increase in baseline pain medications within 4 weeks of the Day 90 visit.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) for Pain | 30 and 90 days
  Scores from daily diaries at 30 and 90 days (analysis will include a comparison of compliance across treatment groups)
Brief Pain (BPI Inventory | 90 days
  The secondary endpoints of this trial are between group comparisons
Daily Sleep Interference Scale (DSIS) | 30 and 90 days
  The secondary endpoints of this trial are between group comparisons
5D-5D-3L | 90 days
  The secondary endpoints of this trial are between group comparisons
Patient Global Impression of Change (PGIC) | 90 days
  The secondary endpoints of this trial are between group comparisons
Depression Anxiety Stress Scales (DASS) | 90 days
  The secondary endpoints of this trial are between group comparisons b
Pain Disability Index (PDI) | 90 days
  The secondary endpoints of this trial are between group comparisons

OTHER OUTCOMES:
Reduction or elimination non-opioid pain medications | 365 Days
  Subjects on Axon Therapy and based on prescribed dosages
Improvement in PDI score | 365 Days
  Proportion of subjects with clinically meaningful change as 10 point improvement, in PDI score 365 days post start of treatment as compared to baseline, subjects on a Axon Therapy
Mean/percent reduction in morphine equivalent daily dose (MEDD) | Day 180 and 365
  Based on prescribed dosages with Axon Treatment Therapy or Gabapentin equivalence for any CMM subjects
Proportion of subjects who discontinue treatment and/or change treatment arms | Day 90
  Proportion of subjects who discontinue treatment and/or change treatment arms
Proportion of subjects in each satisfaction category at Day 180 and 365 (Subjects on Axon Therapy). | Day 180 and Day 365
  Proportion of subjects in each satisfaction category at Day 180 and 365 (Subjects on Axon Therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Joe Milkovits, Study Director — NeuraLace Medical
Locations (3):
- United States (3):
  - National Spine and Pain Centers, Shrewsbury, New Jersey
  - Carolinas Pain Institute, Winston-Salem, North Carolina
  - SC Pain and Spine Specialists (Crescent Moon Research Corp), Murrells Inlet, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kapural L, Patel J, Rosenberg JC, Li S, Amirdelfan K, Bedder M. Efficacy and Safety of Magnetic Peripheral Nerve Stimulation for Treatment of Neuropathic Pain; One Year Follow Up of Long-Term Outcomes. J Pain Res. 2025 Aug 30;18:4471-4481. doi: 10.2147/JPR.S538263. eCollection 2025. PMID 40918409